CLINICAL TRIAL: NCT00795106
Title: Double-blinded, Cross-over Randomized Controlled Trial to Evaluate the Efficacy of Topical Capsaicin to Reduce Pain and Improve Health-related Quality of Life in Adults With Chronic Myofascial Neck Pain
Brief Title: Trial to Evaluate the Efficacy of Topical Capsaicin to Reduce Pain and Improve Health-related Quality of Life in Adults With Chronic Myofascial Neck Pain
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty finding a monitor
Sponsor: Stamford Hospital (Other)
Responsible Party: Marc Brodsky, Medical Director, Center for Integrative Medicine and Wellness at Stamford Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-1014.01
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Myofascial Pain Syndrome
Keywords: Capsaicin; hydrogel; myofascial pain syndrome; neck pain
MeSH Terms: conditions — Myofascial Pain Syndromes; Neck Pain | interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capsaicin patch (Active Comparator): Patches will contain capsaicin 0.1% (500 mcg)
  Interventions: Drug: Capsaicin
- Placebo patch (Placebo Comparator): Placebo hydrogel patches will be 2.5 cm in diameter with a breathable cloth backing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Capsaicin — Each group will undergo two 4-week treatment arms separated by a 4-week wash-out period. Participants will apply 1 hydrogel patch on both the right-sided and left-sided neck and shoulder girdle on the skin overlying a myofascial trigger point. No more than 2 patches will be used on each subject per treatment. During each 24-hour period, the patches will be placed on the skin for 12 hours and will be removed for 12 hours. Placebo hydrogel patches will be 2.5 cm in diameter with a breathable cloth backing. The experimental patches will be identical to placebo patches except will contain capsaicin 0.1% (500 mcg).
  Arms: Capsaicin patch
Drug: Placebo — Each group will undergo two 4-week treatment arms separated by a 4-week wash-out period. Participants will apply 1 hydrogel patch on both the right-sided and left-sided neck and shoulder girdle on the skin overlying a myofascial trigger point. No more than 2 patches will be used on each subject per treatment. During each 24-hour period, the patches will be placed on the skin for 12 hours and will be removed for 12 hours. Placebo hydrogel patches will be 2.5 cm in diameter with a breathable cloth backing. The experimental patches will be identical to placebo patches except will contain capsaicin 0.1% (500 mcg).
  Arms: Placebo patch

SUMMARY:
Chronic neck pain is a common condition that can negatively impact quality of life. Substance P is one of the chemicals in the body that can transmit pain signals from overloaded neck muscles to the brain. Topical capsaicin blocks the action of Substance P by releasing, and subsequently depleting the body's store of Substance P in the nerves. Topical capsaicin has been reported to be an effective therapy for a number of persistent pain conditions including diabetic neuropathy, post-herpetic neuralgia, osteoarthritis, rheumatoid arthritis, and post-mastectomy pain. This study will evaluate the efficacy of topical capsaicin to reduce pain and improve health-related quality of life in adults with chronic muscular neck pain.

DETAILED DESCRIPTION:
The study will employ a double blinded randomized controlled cross-over trial design. A total of 60 patients aged 18-65 with at least 3 months of myofascial neck pain will be recruited to participate in the study. The participants will be randomized into two groups. Each group will undergo two 4-week treatment arms separated by a 4-week wash-out period. Participants will apply a topical gel patch 12 hours each day overlying painful areas in the neck and shoulder girdle for each 4-week period. The topical gel patch used in each arm of the study will be identical except the placebo will not contain the active ingredient, 0.1% capsaicin. Both topical gel patches will be supplied by Caleb Pharmaceuticals. Each participant will complete 3 surveys at baseline and after each 4-week treatment arm: 1) McGill Pain Scale, 2) visual analog scale, and 3) Short Form 36 (general quality of life data). Paired T-tests will be used to evaluate for statistically significant changes between treatment with the control gel versus the active ingredient gel containing the capsaicin.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Speak, read, and write English who have greater than 3 month duration of myofascial neck pain.

Exclusion Criteria:

* Patients who have used capsaicin in the last 4 months and patients with allergy to capsaicin
* Rash/infection overlying neck and shoulder girdle area
* Radiculopathy or structural abnormalities in the area being treated
* Unstable underlying diseases such as cardiovascular, hepatic, renal and CNS disorders will be excluded from the study
* Pregnant or breast-feeding women will not be allowed to participate in the study, and women of child bearing age will be using an effective method of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 1 month

SECONDARY OUTCOMES:
Quality of life | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Marc Brodsky, MD, Principal Investigator — Stamford Hospital
Locations (1):
- Stamford Hospital, Stamford, Connecticut, United States